CLINICAL TRIAL: NCT02934776
Title: Prospective Cohort Study of the Ability of MRI/DTI to Diagnose Prostate Cancer in Men Undergoing Prostate MRI
Brief Title: Prospective Cohort Study of the Ability of MRI/DTI to Diagnose Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rabin Medical Center (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, david margel, Staff Uro-Oncologist, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0357-16-RMC
Record Dates: First submitted 2016-10-11; First posted 2016-10-17 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Magnetic Resonance Imaging
Keywords: DTI; prostate cancer; MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DTI acquisition (Experimental): Addition of up to 10 minutes in MRI machine purpose of acquiring additional DTI images
  Interventions: Device: MRI machine

INTERVENTIONS:
Device: MRI machine — The Philips Ingenia 3.0T is an MRI machine intended to be used by specialist radiologists in the hospital. It is able to acquire high quality images of wide variety of organs. For imaging the prostate, T2-weighted turbo spin-echo images are normally obtained in three orthogonal planes (axial, sagittal and coronal). This device is been clinically used in the MRI department in Belinson hospital.
  Other Names: Ingenia 3.0T

SUMMARY:
The purpose of this study is to examine if investigators can improve diagnosis of prostate cancer by using MRI/DTI?

DETAILED DESCRIPTION:
This is a prospective cohort study of the ability of MRI/DTI to diagnose prostate cancer in men undergoing prostate MRI.

Study design: Male adults who are scheduled to undergo MRI of the prostate, for clinical reasons, will be subjected to additional 10 minutes of image acquisition inside the MRI machine. The added MRI/DTI acquisition does not involve injection of additional contrast material. Investigators will compare between ability of the full mp-MRI images to diagnose prostate cancer to that of the MRI/DTI images

ELIGIBILITY:
Inclusion Criteria:

1. Men who are scheduled to undergo MRI of the prostate at the Department of Imaging, in Beilinson Hospital, Rabin Medical Center
2. Age 18-90.
3. Men who are willing and able to sign an informed consent form.

Exclusion Criteria:

1) Men who cannot complete the full acquisition of the MRI and the MRI/DTI image sequences for any reason.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Compare between number of prostate cancer diagnosed by mpMRI to the ones diagnosed by MRI/DTI | 1 year

SECONDARY OUTCOMES:
Compare the correlation of MRI/DTI parameters with prostate cancer diagnosis to the ones measured by mpMRI (ADC, and diffusion weighted images). | 1 year
Compare between MRI/DTI and MRI ability to identify low-grade and high-grade prostate cancer | 1 year
Compare between MRI/DTI and MRI in their ability to estimate tumor size. | 1 year
Compare between MRI/DTI and MRI in PiRAD grading | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided